CLINICAL TRIAL: NCT05824663
Title: A Phase 1 Open-label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Anti-tumor Activity of HBM1020 in Subjects With Advanced Solid Tumors
Brief Title: A Study Evaluating the Safety, Tolerance and Anti-tumor Activity of HBM1020 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Harbour BioMed US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1020.1
Record Dates: First submitted 2023-03-24; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: Advanced Solid Tumor
Keywords: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HBM1020 (Experimental): HBM1020 is a recombinant fully human anti-B7H7 monoclonal antibody
  Interventions: Drug: HBM1020

INTERVENTIONS:
Drug: HBM1020 — Intravenous (IV) Administrations on Days 1 of each 21-day treatment cycle.

SUMMARY:
This is a study to evaluate the safety and tolerability of the study drug HBM1020 which contains two parts. Part 1 will enroll solid tumor participants and Part 2 will enroll renal cell carcinoma (RCC) and colorectal adenocarcinoma (CRC).

DETAILED DESCRIPTION:
This is a study to evaluate the safety and tolerability of the study drug HBM1020, and to determine the maximum tolerated dose and/or recommended Phase 2 study dose of HBM1020. The study will also look at the anti-tumor activity of HBM1020.The study consists of 2 parts. In Part 1, patients are enrolled into different cohort doses in order to identify the appropriate recommended phase 2 dose (RP2D) or maximum tolerated dose (MTD). In Part 2, participants with metastatic/unresectable RCC, CRC will receive the MTD and/or RP2D established in Part 1 of the study. In Part 1 and Part 2, participants will be administered treatment every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Willingness to sign a written informed consent document.
2. Male or female subject aged ≥18 years old at the time of screening.
3. Histologically or cytologically confirmed advanced solid tumors or recurrent and progressed since last antitumor therapy for which no alternative, curative standard therapy exists.
4. Adequate organ and bone marrow function.

Exclusion Criteria:

1. Prior used anti-B7H7 monoclonal antibodies (mAb) or anti-KIR3DL3 monoclonal antibodies (mAb).
2. Any systemic anti-cancer therapy within 4 weeks prior to first dose of investigational medicinal product (IMP), or immunosuppressive medications within 2 weeks before the first dose of investigational medicinal product (IMP).
3. Not yet recovered from surgery or (immune-related) toxicity related with previous treatment.
4. With clinically significant congenital or acquired cardiovascular diseases.
5. With severe or uncontrolled systemic diseases, including uncontrolled hypertension, uncontrolled diabetes mellitus, active bleeding diatheses, or active infection including hepatitis B, hepatitis C, autoimmune disease and human immunodeficiency virus.
6. Presence of other active invasive cancers other than the one treated in this study within 5 years prior to screening, except appropriately treated basal cell carcinoma of the skin, or in situ carcinoma of uterine cervix, or other local tumors considered cured by local treatment.
7. Major surgery (excluding placement of vascular access) within 4 weeks of first dose of study drug.
8. Previously untreated brain metastases.
9. Pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-05 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with dose-limiting toxicity (DLT) | From Day 1 until disease progression or Day 21, whichever comes first.
  Number of subjects who experience dose-limiting toxicity (DLT) events during 21 days

SECONDARY OUTCOMES:
Adverse events (AEs) | From the date of informed consent until safety follow-up Day 90.
  According to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 (including vital signs, physical examinations, and abnormal laboratory parameters).
Objective response rate (ORR) | Up to 2 years or until progressive disease, unacceptable toxicity, subject withdraw consent or investigator's decision, whichever occurs first.
  The proportion of subjects with best overall response of complete response (CR) or partial response (PR) per RECIST 1.1
Duration of response | Up to 2 years or until progressive disease, unacceptable toxicity, subject withdraw consent or investigator's decision, whichever occurs first.
  The time interval from first occurrence of a documented objective response to the time of disease progression as determined by the Investigator using RECIST 1.1 or death from any cause, whichever comes first
Disease control rate | Up to 2 years or until progressive disease, unacceptable toxicity, subject withdraw consent or investigator's decision, whichever occurs first.
  The proportion of subjects with a best overall response of CR, PR, or stable disease (SD)
Duration of disease control | Up to 2 years or until progressive disease, unacceptable toxicity, subject withdraw consent or investigator's decision, whichever occurs first
  The time from the date of start of treatment to the date of disease progression or death for subjects who had CR or PR or SD during treatment
Tumor shrinkage (The percentage of patients with tumor shrinkage) | Up to 2 years or until progressive disease, unacceptable toxicity, subject withdraw consent or investigator's decision, whichever occurs first.
  The greatest tumor shrinkage achieved at any follow-up assessment. Measured by radiological (computed tomography [CT]/Magnetic Resonance Imaging [MRI]) scanning until documented radiographic disease progression according to RECIST 1.1, or loss of clinical benefit after disease progression according to RECIST 1.1
Maximum serum concentration (Cmax) | Up to 90 days after end of treatment.
  Maximum serum concentration
Time to reach maximum serum concentration (Tmax) | Up to 90 days after end of treatment.
  Time to reach maximum serum concentration
Area under the serum concentration versus time curve from time zero to the dosing interval tau (AUC0-tau) | Up to 90 days after end of treatment.
  area under the serum concentration versus time curve from time zero to the dosing interval tau

IPD SHARING:
Plan to Share IPD: No